CLINICAL TRIAL: NCT01826513
Title: AutoSet for Her Clinical Trial Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Collaborators: The University of Western Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MA13245678
Record Dates: First submitted 2013-04-01; First posted 2013-04-08 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Efficacy; Subjective feedback; Preference
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Unblinded Investigational Arm (Experimental): Participants participated in an unblinded investigational phase of the trial prior to, and separate from, the single-blind cross-over phase of the trial. Data was collected from the his phase to aid the final development of the algorithm before proceeding to algorithm validation (ie. cross-over phase).
  Interventions: Device: Modified AutoSet algorithm
- Standard AutoSet algorithm (Active Comparator): Participants first received therapy with the Standard AutoSet algorithm for one night, and then received therapy with the Modified AutoSet algorithm (an AutoSet device with an algorithm developed for sleep breathing parameters specific to females) the following night.
  Interventions: Device: Standard AutoSet algorithm; Device: Modified AutoSet algorithm
- Modified AutoSet algorithm (Experimental): Participants first received therapy with the Modified AutoSet algorithm (an AutoSet device with an algorithm developed for sleep breathing parameters specific to females) for one night, and then received therapy with the standard AutoSet algorithm the following night.
  Interventions: Device: Standard AutoSet algorithm; Device: Modified AutoSet algorithm

INTERVENTIONS:
Device: Standard AutoSet algorithm — An AutoSet device with a standard algorithm developed for sleep breathing parameters that are specific to a particular gender.
  Arms: Modified AutoSet algorithm; Standard AutoSet algorithm
Device: Modified AutoSet algorithm — An AutoSet device with an algorithm developed for sleep breathing parameters specific to females.
  Other Names: AutoSet for Her

SUMMARY:
The purpose of this study is to assess the efficacy and user preference of the Newport AutoSet for Her in female obstructive sleep apnea (OSA) patients.

Efficacy will be evaluated by comparing the apnea and hypopnea index (AHI) and oxygen desaturation index (ODI) of the Newport AutoSet for Her algorithm to a standard algorithm.

User preference will be evaluated by subjective feedback relating to comfort, ease of falling asleep, sleep disturbance and feeling of being refreshed.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal females aged ≥ 18 years
* Current positive airway pressure (PAP)(CPAP or APAP) therapy user with 'current' defined as on PAP therapy for at least 1 month prior to study entry
* Diagnostic PSG available
* Diagnosis of mild-moderate OSA (AHI ≤ 30)
* Participants willing and able to give written informed consent

Exclusion Criteria:

* Participants currently using Bi-level PAP
* Participants currently using supplemental oxygen
* Participants who are pregnant
* Subjects who have a pre existing lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury)
* Participants who the researcher believes are unsuitable for inclusion because either:

  * they do not comprehend English
  * they are unable to provide written informed consent
  * they are physically unable to comply with the protocol

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Eastwood, MBBS FRACP, Principal Investigator — Centre for Sleep Science, University of Western Australia; David Hillman, MBBS FRACP, Principal Investigator — West Australian Sleep Disorders Reserach Institute
Locations (1):
- West Australian Sleep Disorders Research Institute, Nedlands, Western Australia, Australia

RESULTS

PARTICIPANT FLOW:
Groups:
- Modified AutoSet Then Standard AutoSet: Participants first received therapy with the Modified AutoSet algorithm (an AutoSet device with an algorithm developed for sleep breathing parameters specific to females) for one night, and then received therapy with the standard AutoSet algorithm the following night.
Period: Overall Study
Arm/Group | Unblinded Investigational Arm | Standard AutoSet Algorithm | Modified AutoSet Then Standard AutoSet
Started | 5 | 10 | 10
Completed | 5 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unblinded Investigational Arm | Standard AutoSet Algorithm | Modified AutoSet Then Standard AutoSet | Total
Number analyzed (Participants) | 5 | 10 | 10 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.60 (7.70) | 44.10 (3.78) | 45.60 (6.13) | 44.85 (5.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 10 | 25
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 5 | 10 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: Apnoea Hypopnoea Index (AHI)
Description: Number of apnoeas and hypopnoeas per hour of sleep
Time Frame: 1 day
Population: Reported results only include data from the blinded cross-over sequence arms (ie. Standard and Modified AutoSet algorithms). Data from the Unblinded Investigational phase of the trial was excluded as this phase was exploratory only to help refine the algorithm, and so, was not intended to be included in the final dataset.
Measure: Mean (Standard Deviation); unit: events/hour
Groups:
- Standard AutoSet Algorithm: Participants completed 1 night receiving therapy with the Standard AutoSet algorithm.
- Modified AutoSet Algorithm: Participants completed 1 night receiving therapy with the Modified AutoSet algorithm.
Arm/Group | Standard AutoSet Algorithm | Modified AutoSet Algorithm
Number analyzed (Participants) | 20 | 20
events/hour | 0.96 (1.40) | 0.91 (0.90)

2. Primary Outcome: Oxygen Desaturation Index (ODI)
Description: Number of oxygen desaturations per hour of sleep
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Standard AutoSet Algorithm | Modified AutoSet Algorithm
Number analyzed (Participants) | 20 | 20
events/hour | 1.92 (1.82) | 2.19 (2.15)

3. Secondary Outcome: Sleep Efficacy
Description: Sleep time divided by total time available for sleep
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total recorded time
Arm/Group | Standard AutoSet Algorithm | Modified AutoSet Algorithm
Number analyzed (Participants) | 20 | 20
percentage of total recorded time | 85.99 (8.55) | 84.14 (9.62)

4. Secondary Outcome: Wake After Sleep Onset Time
Description: Time awake in minutes after initial sleep onset
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Standard AutoSet Algorithm | Modified AutoSet Algorithm
Number analyzed (Participants) | 20 | 20
minutes | 47.52 (34.57) | 57.42 (43.31)

5. Secondary Outcome: Time Taken to Fall Asleep
Description: Time in minutes taken to fall alseep
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Standard AutoSet Algorithm | Modified AutoSet Algorithm
Number analyzed (Participants) | 20 | 20
minutes | 16.52 (19.58) | 16.25 (12.70)

6. Secondary Outcome: Number of Spontaneous Arousals
Description: Number of spontaneous arousals occurring over the entire total sleep time
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Spontaneous Arousals
Arm/Group | Standard AutoSet Algorithm | Modified AutoSet Algorithm
Number analyzed (Participants) | 20 | 20
Spontaneous Arousals | 85.55 (40.88) | 81.40 (33.91)

7. Secondary Outcome: Number of Hypopnoeas
Description: Total number of hypopnoeas occurring in the total sleep time
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hypopneas
Arm/Group | Standard AutoSet Algorithm | Modified AutoSet Algorithm
Number analyzed (Participants) | 20 | 20
Hypopneas | 1.45 (2.33) | 2.00 (3.42)

8. Secondary Outcome: Number of Obstructive Apnoeas
Description: Total number of obstructive apnoeas occurring in the total sleep time
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Obstructive Apnoeas
Arm/Group | Standard AutoSet Algorithm | Modified AutoSet Algorithm
Number analyzed (Participants) | 20 | 20
Obstructive Apnoeas | 1.30 (4.44) | 0.80 (1.36)

9. Secondary Outcome: Number of Central Apnoeas
Description: Total number of central apnoeas occurring in the total sleep time
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Central Apnoeas
Arm/Group | Standard AutoSet Algorithm | Modified AutoSet Algorithm
Number analyzed (Participants) | 20 | 20
Central Apnoeas | 3.55 (7.45) | 3.00 (3.78)

10. Secondary Outcome: Oxygen Saturation
Description: Oxygen saturation recorded in the total sleep time
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage SpO2
Arm/Group | Standard AutoSet Algorithm | Modified AutoSet Algorithm
Number analyzed (Participants) | 20 | 20
percentage SpO2 | 96.56 (0.78) | 96.31 (0.81)

11. Secondary Outcome: Percentage of Total Sleep Time Spent in Each Sleep Stage
Description: Percentage of total sleep time spent in each sleep stage (ie. N1, N2, N3 and REM)
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total sleep time
Arm/Group | Standard AutoSet Algorithm | Modified AutoSet Algorithm
Number analyzed (Participants) | 20 | 20
percentage of total sleep time
  Time spent in N1 Sleep | 6.05 (4.63) | 6.20 (3.33)
  Time spent in N2 Sleep | 51.28 (12.91) | 49.44 (12.01)
  Time spent in N3 Sleep | 24.83 (11.58) | 24.60 (10.77)
  Time spent in REM Sleep | 17.93 (11.05) | 19.77 (7.54)

12. Secondary Outcome: Number of Respiratory Event Related Arousals
Description: Total number of respiratory event related arousals over the entire sleep period
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Respiratory-Event Related Arousals
Arm/Group | Standard AutoSet Algorithm | Modified AutoSet Algorithm
Number analyzed (Participants) | 20 | 20
Respiratory-Event Related Arousals | 2.60 (3.32) | 1.30 (1.84)

ADVERSE EVENTS:
Arm/Group | Unblinded Investigational Arm | Standard AutoSet Algorithm | Modified AutoSet Then Standard AutoSet
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/5 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has the right to

* review
* provide comments (site is not bound to follow them)
* request delay of publication for no more than 120 days to allow for securing of IP
* request the removal of specified confidential information

within 40 days of the proposed publication being released to those not bound by confidentiality obligations.